CLINICAL TRIAL: NCT06926361
Title: Effects of Mindfulness-based Interventions on Improving Teacher Wellbeing and Teaching Outcomes
Brief Title: Effects of Mindfulness-based Interventions on Improving Teacher Wellbeing and Teaching Outcomes: A Multi-site, Mixed-methods Randomized Controlled Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The University of Hong Kong (Other); University of Macau (Other)
Responsible Party: Principal Investigator, Jennifer Yee Man Tang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SBRE-24-0445
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Mental Health; Teaching Skills
Keywords: Mindfulness; Teachers; School; Professional development
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mindfulness for Life (Experimental): MBCT-L is an 8-week program consisting of mindfulness practices and cognitive-behavioral techniques with 8 sessions (2 hours and 15 minutes per session) and one-day retreat that can provide participants with an extended period to deepen their personal mindfulness practices.
  Interventions: Behavioral: Mindfulness for Life
- Positive education training (Active Comparator): Positive Education program is an 8-week course consisting of theories and activities of positive psychology to enhance teachers' skills to support students' learning and wellbeing using a strength-based approach.
  Interventions: Behavioral: Positive education training

INTERVENTIONS:
Behavioral: Mindfulness for Life — Behavioral: Mindfulness for Life (MBCT-L) MBCT-L is an 8-week program consisting of mindfulness practices and cognitive-behavioral techniques with 8 sessions (2 hours and 15 minutes per session) and one-day retreat that can provide participants with an extended period to deepen their personal mindfulness practices.
  Arms: Mindfulness for Life
Behavioral: Positive education training — Positive Education program is an 8-week course consisting of theories and activities of positive psychology to enhance teachers' skills to support students' learning and wellbeing using a strength-based approach.
  Arms: Positive education training

SUMMARY:
This study aims to evaluate the effectiveness of MBCT-L among Chinese teachers on their mental well-being and teaching outcomes and explore the mechanisms of how mindfulness practice brings these benefits. The study is a multi-site, mixed-methods randomized controlled trial including 160 teachers.

ELIGIBILITY:
Inclusion Criteria:

1. Teachers aged 21-65 years;
2. Teachers currently working in a school; and
3. Teachers willing to commit time for the 8-week course.

Exclusion Criteria:

1. Teachers previously joined a related group mindfulness-based intervention, such as mindfulness-based cognitive therapy (MBCT), mindfulness-based stress reduction (MBSR), Mindfulness - Finding Peace in a Frantic World (FPFW); or
2. Teachers who are mentally unstable or having active suicidal risk.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Teaching efficacy | Baseline, 9 weeks, and 3 months post-intervention
  The Teachers' Sense of Efficacy Scale-Short Form (TSES-SF). Participants will rate their responses on a 9-point Likert scale ranging from 1 (nothing) to 9 (a great deal). A higher total score indicates a higher sense of teaching efficacy of teachers.
Teaching practices | Baseline, 9 weeks, and 3 months post-intervention
  The Classroom Strategies Scale-Teacher Form (CSS-T). Participants will rate their frequency of using a specific strategy in two domains on a 7-point Likert scale from 1 (never used) to 7 (always used). Higher scores indicate teachers use specific strategies more frequently.
Classroom climate | Baseline, 9 weeks, and 3 months post-intervention
  Three subscales of Delaware School Climate Scale-Teacher/Staff (DSCS-T/S): Student-Student Relations, Student Engagement, and Clarity of Expectations. It uses a 4-point Likert scale from 1 (disagree a lot) to 4 (agree a lot). A higher total score indicates a better classroom climate.

SECONDARY OUTCOMES:
Stress | Baseline, 9 weeks, and 3 months post-intervention
  The Perceived Stress Scale. Participates rate their stress on a 5-point Likert scale ranging from 0 (never) to 4 (very often). A higher total score indicates higher stress levels.
Anxiety | Baseline, 9 weeks, and 3 months post-intervention
  Generalized Anxiety Disorder Assessment (GAD-7). The items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day) over the past two weeks. A higher total score indicates a higher level of anxiety.
Depression | Baseline, 9 weeks, and 3 months post-intervention
  The Patient Health Questionnaire-9 (PHQ-9). The items are rated on a 4-point Likert scale ranging from 0 (not at all) to 3 (nearly every day) over the past two weeks. A higher total score indicates higher depressive symptoms.
Burnout | Baseline, 9 weeks, and 3 months post-intervention
  Maslach Burnout Inventory - Educators Survey (MBI-ES). Participants report scores on a 7-point Likert scale ranging from 0 (never) to 6 (every day). A higher total score indicates a higher level of burnout.

OTHER OUTCOMES:
Trait mindfulness | Baseline, 9 weeks, and 3 months post-intervention
  The Five-Facet Mindfulness Questionnaire (FFMQ-15). Participants give ratings on a 5-point Likert scale from 1 (never or very rarely true) to 5 (very often or always true). A higher total score means a higher level of trait mindfulness.
Emotion regulation | Baseline, 9 weeks, and 3 months post-intervention
  The Emotion Regulation Questionnaire (ERQ). Participants will rate their responses on a 7-point Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree). A higher total score in each subscale indicates a higher tendency of using the specific emotion regulation strategy.